CLINICAL TRIAL: NCT06965907
Title: Immediate Effect of Kinesio Taping on Two-Point Discrimination, Fine Motor Skills, Grip Strength and Reaction Time on Computer Users
Brief Title: Kinesiotaping on Hand Function in Computer Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Çiçek Günday, Asst. Prof., Istinye University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29032002
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Computer-user Training
Keywords: kinesiotaping; sensation; dexterity; reaction time; athletic tape

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping group (Experimental)
  Interventions: Other: Kinesio Taping
- Sham Kinesio Taping group (Sham Comparator)
  Interventions: Other: Sham Taping

INTERVENTIONS:
Other: Kinesio Taping — The participant will be seated upright in a chair with the elbow flexed at 90 degrees. The forearm under examination will be placed in a pronated position, and the wrist will be maintained in a neutral position. I-shaped kinesio taping will be applied as described by Mohammadi et al. Prior to taping, the extensor surface will be cleaned using a cotton swab moistened with alcohol. The tape length will be measured from a point 2 cm distal to the lateral epicondyle to the radial styloid process. Each end of the tape will be 2 cm in length (totaling 4 cm for both ends). To achieve 35% tension, the following formula will be used: (L - 4) / 1.35 + 4. In this formula, L represents the total length of the tape, 4 is the combined length of the two tape ends, and 1.35 corresponds to the factor required to achieve the desired 35% tension.
  Arms: Kinesio Taping group
Other: Sham Taping — The participant will be seated in a chair with the forearm resting comfortably. The tape will be applied to the middle of the forearm without any tension. The taping will be performed from the medial to the lateral direction.
  Arms: Sham Kinesio Taping group

SUMMARY:
This study aims to investigate whether kinesio taping contributes to improved hand function in individuals who frequently use computers. The effectiveness of kinesio taping will be compared to sham taping in order to determine its impact. Participants will be randomly assigned to one of two groups: a kinesio taping group or a sham taping group. Taping will be applied to the forearm. Functional assessments will be conducted at three time points: prior to taping, immediately after taping, and 30 minutes post-taping. The following evaluations will be performed:

* Two-point discrimination test to assess touch sensitivity
* Purdue Pegboard test to evaluate fine motor skills
* Grip strength test using a hand dynamometer
* Visual reaction time test utilizing a light-based device All procedures will be completed in a single study session.

ELIGIBILITY:
Inclusion Criteria:

* Participants must use a computer ≥ 2 hours per day.
* Participants must be between the ages of 18 and 50.
* If the participants are employed, they must not have changed professions in the last 6 months.
* If the participants are students, their student status must have been ongoing for at least 6 months.

Exclusion Criteria:

* A diagnosed history of neuropathy or common diseases associated with peripheral neuropathy.
* Diagnosed musculoskeletal disorders related to the neck and upper extremities.
* Presence of symptoms suggestive of nerve entrapment.
* Having a condition that prevents the application of physical tests (e.g., limited range of joint motion, deformities, fractures, arthritis, etc.).
* Allergic reaction to kinesiology tape.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Two-point Discrimination | Day 1
  This test measures an individual's ability to perceive two closely spaced points touching the skin simultaneously, reflecting tactile spatial acuity. During the evaluation, the contact points will initially be set 14 mm apart, with the distance reduced by 1 mm at each step. Adjustments will continue until the participant can no longer distinguish two separate points. The final distance at which two points are still perceived as distinct will be recorded.
Fine Motor Skills | Day 1
  Purdue Pegboard Test will be used. The participant will be seated at a table with the pegboard placed directly in front of them. The test consists of four tasks:
  * Dominant Hand Task: The participant will insert as many pegs as possible into the holes using the dominant hand within 30 seconds.
  * Non-Dominant Hand Task: The same procedure will be repeated using the non-dominant hand.
  * Both Hands Task: Pegs will be inserted into the holes in pairs using both hands simultaneously over a 30-second period.
  * Assembly Task: Using both hands, the participant will assemble a sequence using pegs, washers, and collars for a duration of 60 seconds.
  The score will be determined by the number of pegs placed or sequences completed within the specified time limits.
Grip Strength | Day 1
  Maximum grip strength will be measured using a JAMAR Hydraulic Hand Dynamometer. The participant will be seated upright with the elbow flexed at 90 degrees, and the forearm and wrist maintained in a neutral position. Participants will be instructed to squeeze the dynamometer with maximum effort for five seconds. Three trials will be conducted, with a 30-second rest period between each attempt. The highest value obtained will be recorded as the maximum grip strength.
Reaction Time | Day 1
  Reaction time will be recorded using the BlazePod Trainer device. BlazePod is a wireless lighting system consisting of LED pods and a control unit. Participants will begin the test in a seated position, placing their hands on the table with palms facing downward and spaced 40 cm apart. The BlazePod will be positioned at the center of the table, 20 cm away from each hand, and will emit random light signals. Participants will be instructed to tap the illuminated pod as quickly as possible upon activation. The test will last for 15 seconds, and the average reaction time of all hits during the activity will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University Physiotherapy and Rehabilitation Application and Research Center (İSÜFİZYOTEM), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No